CLINICAL TRIAL: NCT06012162
Title: Long-read Genome Sequencing and Risk Stratification of Myocardial Ischemia in Patients With Heart Transplantation
Brief Title: Genomics in Heart Transplants
Status: Not yet recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: Genomics in HTx
Record Dates: First submitted 2023-04-04; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Heart Transplantation
Keywords: heart transplantation; long-read genomics; risk stratification; myocardial ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of blood samples through clinical routine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional analysis of 200 heart transplant recipients, combining in-depth phenotyping and risk factor assessment (cardiac MRI, coronary angiogram with OCT, cardiorespiratory exercise tests, exogenic factors like nutrition, smoking, lipid profile) with short-read whole-genome sequencing to elucidate the interplay of established PRS from the literature and exogenic risk factors with respect to HTx outcomes will be carried out.

Besides that, a long-read whole-genome sequencing of 100 newly transplanted recipients and their corresponding donors and extend latest bioinformatics methods developed by the study to analyze long-read data will be performed. This will enable a comprehensive and integrated analysis of structural variants, polygenic risk, high-penetrance variant genotypes, immunogenetic (major and minor histocompatibility), and individual lifestyle risk factors in a unique donor-recipient cohort, elucidating the extent of within-cohort variability and cross-correlations between the considered potential risk factors and an exploratory analysis of the utility of genetic risk scores in light of the study results will be carried out.

DETAILED DESCRIPTION:
Background: Heart transplantation (HTx) is the treatment of choice for patients with end-stage heart failure who remain symptomatic despite optimal medical therapy. Even with best-practice follow-up care, one out of eight HTx patients eventually die of ischemic cardiomyopathy and recurrent acute myocardial infarction (AMI). Classical risk factors like the recipient indication for heart transplantation explain a fraction of adverse outcomes, but no conventional risk factor alone satisfactorily predicts the probability of cardiac allograft vasculopathy (CAV) or recurrent AMI in HTx patients; in addition, the underlying pathomechanisms are poorly understood.

Therefore, there is an urgent need for an improved understanding of the factors contributing to recurrent myocardial ischemia in HTx patients. Recent large-scale studies of the genetic architecture of coronary artery disease in the general population indicate that polygenic risk scores (PRS) explain more disease risk than any single non-genetic risk factor, but, due to a lack of longitudinal follow-up studies with deep phenotyping, PRS have not yet been widely adopted in clinical practice. Furthermore, current genetic studies are based on microarrays or short-read sequencing, severely limiting their ability to characterize the effect of complex or structural genetic variation, in the whole human genome as well as in key loci of potential importance for HTx outcomes, affecting, e.g., lipid metabolism (e.g. LPA) and immunogenetic compatibility (e.g. the major histocompatibility complex).

In summary, there is presently no study leveraging the improved ability to resolve human genomes with long-read sequencing technologies in a deeply phenotyped cohort for an improved understanding of recurring myocardial ischemia.

Study design and aims: In an innovative three-component study design, comprehensive phenotyping with the latest long-read sequencing technology and algorithmic advances in computational genomics to elucidate the interplay of genetic and non-genetic risk factors of myocardial ischemia in HTx patients at unprecedented resolution and pave the way towards detailed risk stratification and tailored treatment, will be combined

Significance and translational potential: By enabling the integrated analysis of structural variants, high-penetrance complex variants, and high-resolution immunogenetics, long-read sequencing will enable improved genetic models of the development of ischemia in HTx patients and contribute to an improved understanding of underlying pathomechanisms. Based on this, the investigators will be able to propose schemes to incorporate integrated risk scores in future clinical trials for personalized treatment stratification.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old undergoing heart transplantation in our centre

Exclusion Criteria:

* < 18 years
* incapable of giving consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing heart transplantation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
rate of Clinically significant ischemia | 5 years
  defined by cardiac allograft vasculopathy (CAV) grade >1 & cardiac magnetic resonance imaging (cMRI)

SECONDARY OUTCOMES:
cardiovascular death | 5 years
  cardiovascular event as primary cause of death
myocardial infarction | 5 years
  Incidence of Type I or II myocardial infarction (assessed by CMR, electrocardiogram, laboratory parameters according to the 4th universal definition of myocardial infarction)
Hospitalisation (w/o allograft rejection) | 5 years
  All-cause hospitalisation with exception of acute allograft rejection
Cardiac allograft vasculopathy (macrocirculatory) | 5 years
  Incidence: Coronary angiogram (+/- optic coherence tomography (OCT))
number of coronary microvascular dysfunction | 5 years
  measured by fractional flow reserve
number of coronary microvascular dysfunction | 5 years
  measured by cardiac magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, Prof., Study Chair — Clinic for Cardiology, Pneumology and Angiology at University Hospital Düsseldorf
Locations (1):
- University-Hospital Düsseldorf Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany